CLINICAL TRIAL: NCT05530083
Title: A Cluster Randomized Trial to Evaluate the Effect of Group Education on Smoking Cessation and Blood Pressure in Smoking Elderly Males With Stage 1 and 2 Hypertension
Brief Title: Group Education Helps Smoking Cessation and Hypertension Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension and the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESHC
Record Dates: First submitted 2022-08-24; First posted 2022-09-07 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Smoking Cessation; Hypertension
Keywords: group education; smoking cessation; blood pressure
MeSH Terms: conditions — Smoking Cessation; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group education (Experimental): The investigators will provide experimental groups with group education of smoking cessation, including lectures in groups of 50 to 100 people and panel discussion in groups of 5 to 10 people.
  Interventions: Behavioral: group education
- conventional smoking cessation management (Other): The investigators will provide control groups with conventional smoking cessation management, including regular follow-up of smoking status and giving advice of smoking cessation.
  Interventions: Behavioral: conventional smoking cessation management

INTERVENTIONS:
Behavioral: group education — Group education is one of strategies and behavioural interventions of smoking cessation. Lectures, group meeting for mutual support, discussion of coping skills and suggestions for prevention relapse can help smokers quit smoking by providing support and encouragement from people in same condition.
  Arms: group education
Behavioral: conventional smoking cessation management — Including regular follow-up of smoking status and giving advice of smoking cessation
  Arms: conventional smoking cessation management

SUMMARY:
Smoking elderly males with stage 1 and 2 hypertension who currently smoked at least one cigarette per day and were willing to quit smoke will be invited to this cluster randomized, controlled, interventional, open clinical trial. The investigators will provide participants with group education of smoking cessation and their blood pressure measured at clinic at the sixth month is the primary endpoint. The investigators aim to explore how group education of smoking cessation effects smoking cessation, hypertension control and cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* signed the informed consent
* aged 65 to 84
* new-onset hypertension or poorly controlled hypertension (140mmHg≤systolic blood pressure<180mmHg and (or) 90mmHg≤ diastolic blood pressure<110mmHg)
* smoked last week and smoked more than 1 cigarette per day on average
* be willing to quit smoking
* can communicate normally and cooperate in blood pressure measurements, finishing questionnaires
* complete interventions and follow-up consistently

Exclusion Criteria:

* home systolic blood pressure<130mmHg and (or) home diastolic blood pressure<80 mmHg
* severe communication difficulties (aphasia, hearing impairment, etc.)
* suffering from mental disorders such as anxiety and depression
* cancer confirmed
* with previous serious cardiovascular events such as acute coronary syndrome, acute left heart failure, stroke or with specific cardiovascular therapeutic device such as pacemakers
* other serious physical illness or illness identified by investigators that unable to participant in study
* using specific non-permitted medication currently

Ages: 65 Years to 84 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-12 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
change of clinic systolic blood pressure from baseline at the sixth month | 6 months

SECONDARY OUTCOMES:
Cardiovascular events (cardiovascular death, stroke,myocardial infarction) | 6 months, 1 year, 2years, 3 years
change of clinical blood pressure and home blood pressure from baseline | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
Hypertension control rate | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
Biochemical smoking cessation rate | 6 months
  CO≤6 ppm
Self-reported 7-days smoking cessation rate | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
Self-reported long-term smoking cessation rate | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
  Participants hadn't smoked for at least one month.
Self-reported average number of cigarettes smoked per day | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
Relapse rate | 6 month
Mini-Mental State Examination score | 6 months
  The cognitive function of participants will be assessed by MMSE. The score of MMSE ranges from 0 (worse) to 30 (better).
FEV1-Pulmonary functions | 6 months
  Forced expiratory volume in 1 second (FEV1) is the volume of air exhaled in the first second during forced exhalation after maximum inspiration.
PEF-Pulmonary functions | 6 months
  Peak expiratory flow (PEF), the maximal flow that can be exhaled when blowing out at a steady rate.
FVC-Pulmonary functions | 6 months
  Forced vital capacity (FVC), is the maximum amount of air that can be exhaled when blowing out as fast as possible.
Fagerstrom Test for Nicotine Dependence score | 6 months
  The score of FTND ranges from 0 to 10. Participants with higher scores have higher degree of tobacco dependence and are less likely to maintain the status of smoking cessation.
Carbon monoxide concentration breathed | 6 months
Adverse events, including nicotine withdrawal symptoms and other adverse events. | 1 month, 2 month, 3 month, 6 month, 1 year, 2 years, 3 years
  Nicotine withdrawal symptoms were quantified using the Minnesota Tobacco Withdrawal Scale (MNWS).

IPD SHARING:
Plan to Share IPD: Undecided